CLINICAL TRIAL: NCT02117232
Title: A Randomized Controlled Trial to Evaluate Effectiveness and Safety of the Colonoscopy With the "Visualization" Balloon
Brief Title: Effectiveness and Safety of the Colonoscopy With "Visualization" Balloon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mercy Medical Center (Other)
Responsible Party: Principal Investigator, Sergey Kantsevoy, Director of Therapeutic Endoscopy Mercy Medical Center, Clinical Professor of Medicine University of Maryland School of Medicine, Mercy Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: VB-001
Record Dates: First submitted 2014-04-11; First posted 2014-04-17 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Colonic Adenomatous Polyps
Keywords: colonoscopy; cecal intubation; carbon dioxide insufflation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Visualization balloon (Experimental): Colonoscopy performed with the use of "Visualization" balloon
  Interventions: Device: Visualization balloon
- Traditional CO2-insufflation colonoscopy (Active Comparator): Traditional colonoscopy performed with CO2 insufflation without "Visualization" balloon
  Interventions: Device: Traditional CO2 insufflation colonoscopy

INTERVENTIONS:
Device: Visualization balloon — The "Visualization" Balloon is a disposable medical device that is used during the advancement of the colonoscope inside the colon. The intended use of the "Visualization" Balloon is to help insertion of the colonoscope into the colon without the aid of gas (air or CO2) insufflation as with standard colonoscopy. The "Visualization" Balloon is inserted through the biopsy channel of the colonoscope prior to the colonoscope introduction into the rectum. The "Visualization" Balloon is an inflatable balloon that opens up the lumen of the gastrointestinal tract, thereby allowing the endoscopist to advance the endoscope inside and to view the gastrointestinal tract through the clear balloon.
  Arms: Visualization balloon
Device: Traditional CO2 insufflation colonoscopy — Traditional colonoscopy performed with CO2 insufflation without "Visualization" balloon
  Arms: Traditional CO2-insufflation colonoscopy

SUMMARY:
Colonoscopy has become the "gold standard" in detection of colonic polyps and colon cancer. However, colonoscopy causes significant abdominal discomfort and abdominal pain during and after the procedure, requiring intravenous sedation and use of analgesics. The discomfort and pain are mostly caused by air insufflation and intubation difficulties during advancement of the colonoscope in order the reach the cecum.

Study Hypothesis: Use of the "Visualization" Balloon will facilitate advancement of the colonoscope and will eliminate the need for colonic distention with the air or CO2, which can shortened the length of the procedure, reduce patient's discomfort and can decrease amount of sedatives and analgesics used during colonoscopy.

DETAILED DESCRIPTION:
The goal of this study is to evaluate effectiveness and safety of a "Visualization" Balloon for performance of colonoscopy.

Our hypothesis is that, use of "Visualization" Balloon will decrease colonic distention, patient's discomfort, use of sedatives and analgetics during procedure and will simplify the performance of colonoscopy resulting in shortening of procedure time and increasing the rate of cecal intubation.

Specific aims of the study:

1. To compare procedure time and effectiveness of the "Visualization" Balloon colonoscopy with traditional CO2-insufflation colonoscopy.
2. To compare safety profiles between traditional CO2-insufflation colonoscopy and colonoscopy using the "Visualization" Balloon.

4 STUDY ENDPOINTS 4.1 Primary Outcome To compare the mean cecal intubation time achieved with "Visualization" Balloon colonoscopy, with the mean cecal intubation time achieved with standard colonoscopy using CO2 insufflation.

4.2 Secondary Outcomes

To compare "Visualization" Balloon colonoscopy with standard CO2-insufflation colonoscopy in regards of:

1. Total amount of carbon dioxide (CO2) gas for colonic insufflation used during the procedure.
2. Ease of colonoscope insertion.
3. The length of the colonoscope when it reaches the cecum. 4 Colonoscope withdrawal time and total procedure time.

5. Cecal intubation rate. 6. Total dosage of analgesics and sedative during procedure. 7. Patient satisfaction: perceived pain and discomfort immediately after the procedure and in 24 hours post procedure.

8. Complications during and after colonoscopy. 9. Polyp detection rate.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is undergoing colonoscopy for colo-rectal cancer screening, polypectomy or for diagnostic workup.
2. Subject is able to understand the risks and benefits of participating in the study and must be willing to sign and date the Informed Consent Form for this study approved by the Institutional Review Board (IRB.)
3. Age from 17 to 90 years.
4. Be willing and able to comply with the requirements of the protocol.
5. Be willing to refrain from participating in any other investigational interventional study while enrolled in this study.
6. Female subjects must have a negative pregnancy test within the last 24 hours timeline and have no intentions of becoming pregnant during participation in the study, or be sterilized.

Exclusion Criteria:

1. Subjects with a history of previous colonic resection.
2. Subjects with uncorrectable bleeding disorders (INR more than 1.5, platelet count less than 50,000).
3. Subjects unwilling or unable to give written consent to participate in the investigation or unable to comply with the requirements of the protocol.
4. Subjects with suspected colonic strictures potentially precluding complete colonoscopy.
5. Subjects who received any experimental drug or device within the previous three months.
6. Female subjects who were pregnant or lactating or were intending to become pregnant during the period of the study, or who would not use an adequate method of contraception (contraceptive pill, intra-uterine device) for the duration of the study.
7. Subjects who possessed any psychological condition, or were under treatment for any condition which, in the opinion of the Investigator and/or consulting physicians(s), would constitute an unwarranted risk.

Ages: 17 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2014-03; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Cecal intubation time | Immediately
  Time required to reach cecum

SECONDARY OUTCOMES:
Length of colonoscope when it reaches cecum | Immediately
  Total length of colonoscope when it reaches cecum
Ease of colonoscope insertion | Immediate
  Easy of colonoscope insertion to cecum
Dose of analgesics and sedatives used | Immediately
  Dose of analgesics and sedatives used during insertion and total dose for the entire procedure
Patient satisfaction | Immediately and in 24 hours
  Patient satisfaction: perceived pain and discomfort immediately after the procedure and in 24 hours post procedure.
Total procedure time | Immediately
  Total time required to complete colonoscopy

OTHER OUTCOMES:
Amount of carbon dioxide used | Immediately
  Total amount of carbon dioxide used during colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Sergey V Kantsevoy, MD, PhD, Principal Investigator — Mercy Medical Center
Locations (1):
- Mercy Medical Center, Baltimore, Maryland, United States